CLINICAL TRIAL: NCT05098548
Title: Impact of Pedal Arch Patency on Outcomes of Endovascular Revascularization Procedures in Patients With Chronic Limb Threatening Ischemia
Brief Title: Pedal Arch Revascularization in Patients With Chronic Limb Threatening Ischemia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Moustafa Farouk, principle investigator, Assiut University
Other Study IDs: PARIPWCLTI
Record Dates: First submitted 2021-10-16; First posted 2021-10-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Critical Ischemia of Foot
MeSH Terms: interventions — Angioplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with Chronic limb threatening ischemia: All patients with Chronic limb threatening ischemia present with one or more of the following:
  1. Rest pain (Rutherford category 4)
  2. Minor tissue loss (Rutherford category 5) admitted to the department of Vascular surgery for Endovascular Intervention with provided written informed consent.
  Interventions: Procedure: angioplasty

INTERVENTIONS:
Procedure: angioplasty — using a balloon to stretch open a narrowed or blocked artery. However, most modern angioplasty procedures also involve inserting a short wire-mesh tube, called a stent, into the artery during the procedure. The stent is left in place permanently to allow blood to flow more freely .

SUMMARY:
Chronic limb threatening ischemia (CLTI) is a major cause of morbidity and mortality worldwide and is characterized by multilevel disease, often involving the tibiopedal vessels . CLTI is an undesirable clinical consequence of peripheral arterial disease (PAD) . It affected ∼8 million people in the USA and affects 12-20% of American people aged more than 65 years. Within 1 year of diagnosis, 25% of those patients progress to a major amputation and the other 25% die due to co-morbid conditions

DETAILED DESCRIPTION:
Revascularization is the cornerstone of Chronic limb threatening ischemia (CLTI) treatment for lower limb preservation . Endovascular revascularization is the favored approach in many centers because of its lower morbidity and mortality than open surgery . In a subset of patients with Chronic limb threatening ischemia, particularly in longstanding type 1 diabetic patients, a predominance of disease involving the pedal vessels can exist with relative sparing of the tibial vessels .The pedal arch describes the connection between the anterior and posterior circulation in the foot, this typically runs from the lateral plantar artery into the dorsalis pedis and represents the final arcade of outflow for the lower extremity vasculature . Secondary or "deep" pedal plantar loops connecting the medial and lateral tarsal arteries to the medial and lateral plantar arteries can also exist . A strong understanding of the pedal arch anatomy and its multiple connections is important for the physician performing not only pedal arch interventions, but tibial interventions as well . Familiarity with the arch anatomy increases procedural success rates in tibial intervention, as it gives the operator another collateral pathway to approach the target occlusion in a retrograde fashion . An intact pedal arch has been associated with improved wound healing, as well as a higher patency rate for bypass grafting and percutaneous interventions for inflow disease . An Angio some-directed revascularization strategy, however, has clearly been shown to improve wound healing and limb salvage rates in both surgical and endovascular series . Pedal arch intervention should therefore be considered in patients with advanced tissue loss, with a goal of restoring inline flow to the corresponding angiosomes, this could mean the difference between a major and minor amputation, as the options for these patients are limited and major amputation rates are high .

ELIGIBILITY:
Inclusion Criteria:

All patients with Chronic limb threatening ischemia present with one or more of the following:

* Rest pain (Rutherford category 4)
* Minor tissue loss (Rutherford category 5) admitted to the department of Vascular surgery for Endovascular Intervention with provided written informed consent.

Exclusion Criteria:

* Patients presented with proved vasculitis.
* Patients with Chronic liver disease if there is prolonged PT.
* Patients with Heart failure if the patient is orthopneic and cannot lay on table for long time).
* Patients with impaired renal function.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The calculation was done using confidence interval 98 % giving a total sample size 28. According to the equation for sample size for prospective study design, prevalence of chronic limb threatening ischemia was 1.3 % of total population attending the Vascular Surgery Department [2]. Raising the sample size will be done up to 35 to compensate for dropout and refusal.
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Patency of the vessel | From December 2021 to April 2022
  Primary patency Which means maintaining vessel patency without restenosis or need for re-intervention .

IPD SHARING:
Plan to Share IPD: No